CLINICAL TRIAL: NCT03811704
Title: Real-time Navigation for Laparoscope Liver Resections Using Fusion 3D Imaging and Indocyanine Green Fluorescence Imaging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201802
Record Dates: First submitted 2018-12-02; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-11

CONDITIONS: Liver Resection
Keywords: three-dimensional reconstruction; fluorescence; indocyanine green; liver resection; navigation surgery
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Hepatectomy procedures were performed under Laparoscopic surgical navigation system and Indocyanine Green guidance.
  Interventions: Device: Laparoscopic surgical navigation system; Drug: Indocyanine Green

INTERVENTIONS:
Device: Laparoscopic surgical navigation system — We will use this navigation system to guide de liver resection.
Drug: Indocyanine Green — ICG was administered 24 hours before the operation or intravenously after clamping the Glissonian sheaths flowing in the cancer-bearing hepatic segment, or directly into the portal branches supplying blood flow to the tumor-bearing hepatic segment, after puncturing of the target segments under intraoperative ultrasonography guidance.

SUMMARY:
The aim of this study was to evaluate the feasibility and efficacy of a novel real-time navigation way for laparoscope liver resection, which was fused images comprising 3D imaging and indocyanine green Fluorescence imaging (fusion IGFI).

DETAILED DESCRIPTION:
During liver resection, surgeons cannot completely view the intraparenchymal structure. Although a fluorescent imaging technique using indocyanine green has recently been developed for hepatobiliary surgery, limitations in its application for real-time navigation persist. A nove augmented reality surgery navigation system (ARSNS) can be combined with indocyanine green Fluorescence imaging to guide the surgery real-time.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years≤ Age ≤70 years
2. Compling with the diagnosis criteria of complex hepatic carcinoma.
3. Primary hepatic carcinoma without intrahepatic or extrahepatic extensive cancer metastasis, the metastatic hepatic carcinoma whose primary focal has been controlled
4. Preoperative liver function is Child - Pugh grade A or B.
5. The patients are volunteered for the study.

Exclusion Criteria:

1. Patients with mental illness.
2. Patients can't tolerate the operation owe to a variety of basic diseases (such as severe cardiopulmonary insufficiency, renal insufficiency, cachexia and blood system diseases, etc.)
3. The patients refused to take part in the study.
4. There are other co-existed malignant tumors.
5. Benign liver diseases.
6. Indocyanine green allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Liver resection navigation success rate | intraoperative
  Whether this technique successfully displayed the pre-resection line during the surgery were recorded.

SECONDARY OUTCOMES:
Postoperative complication rate | 3 months
  The Postoperative complications were recorded.
Operative outcomes | intraoperative
  Operative outcomes such as operative time, estimated blood loss and blood transfusion were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chihua Fang, M.D.;Ph.D, Study Director — China, Guangdong Zhujiang Hospital of The Southern Medical University
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhu W, Zeng X, Hu H, Xiang N, Zeng N, Wen S, Tian J, Yang J, Fang C. Perioperative and Disease-Free Survival Outcomes after Hepatectomy for Centrally Located Hepatocellular Carcinoma Guided by Augmented Reality and Indocyanine Green Fluorescence Imaging: A Single-Center Experience. J Am Coll Surg. 2023 Feb 1;236(2):328-337. doi: 10.1097/XCS.0000000000000472. Epub 2022 Nov 8. PMID 36648260